CLINICAL TRIAL: NCT04109989
Title: Clinical Assessment - HominisTM Surgical System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memic Innovative Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MEMIC-5083
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HominisTM Surgical System (Experimental): Gynecological surgical procedure will be performed with the HominisTM Surgical System
  Interventions: Device: HominisTM Surgical System

INTERVENTIONS:
Device: HominisTM Surgical System — Trans-vaginal gynecological procedures

SUMMARY:
A clinical research study designed to assess the HominisTM Surgical System in gynecological procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Female above 18 years of age inclusive.
2. Able to provide written informed consent.
3. Eligible for Total Transvaginal Laparoscopic Hysterectomy with Salpingo-Oophorectomy or Transvaginal Laparoscopic Hysterectomy with Salpingectomy and have an appropriate indication to go through this surgery.
4. Willing to undergo laparoscopic transvaginal procedure by Memic HominisTM Surgical System.
5. Fit for robotic-assisted transvaginal surgery based on surgeon discretion.
6. Can undergo general anesthesia per anesthesiologist assessment.

Exclusion Criteria:

1. Women with anatomical hazard for laparoscopy and/or vaginal and/or pouch of Douglas access (such as diagnosis of Crohn's disease, active Pelvic inflammatory disease (PID), active diverticulitis, sever peritoneal adhesions, frozen pelvis, obliterated vagina or sever recto-vaginal endometriosis).
2. Women after pelvic radiation.
3. Women diagnosed with active intra-abdominal malignancy.
4. Women with general condition or illness incompatible for surgery.
5. Women who are pregnant.
6. Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The device is intended for Vaginal procedures
Enrollment: 50 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion | Intra Operative
  Rate of conversion to open or laparoscopic approach

SECONDARY OUTCOMES:
Intra-operative & post-operative procedural outcomes | Intra-operative and six weeks post procedure
  Intra-operative & post-operative complications
Intra-operative & post-operative procedural outcomes | Intra-operative & six weeks post procedure
  adverse events (AE and SAE)
Intra-operative & post-operative procedural outcomes | Intra-operative & six weeks post procedure
  Bladder injury rate
Intra-operative & post-operative procedural outcomes | Intra-operative & six weeks post procedure
  Rectal injury rate
Intra-operative procedural outcomes | Intra-operative
  Operative time
Intra-operative & post-operative procedural outcomes | Intra-operative & six weeks post procedure
  Transfusion rate
Intra-operative procedural outcomes | Intra-operative
  Conversion rate (to laparotomy, laparoscopy, other ports used in addition to vaginal and umbilical port).
Intra-operative & post-operative procedural outcomes | Intra-operative & six weeks post procedure
  Mortality
Post-operative procedural outcomes | Six weeks post procedure
  Length of hospital stay
Post-operative procedural outcomes | Six weeks post procedure
  Re-admission rate
Post-operative procedural outcomes | Six weeks post procedure
  Re-operation rate
Vaginal tissue healing | Six weeks post procedure
  Vaginal tissue healing will be assessed

CONTACTS AND LOCATIONS:
Locations (2):
- Imelda Hospital, Bonheiden, Belgium
- Rambam Hospital, Haifa, Israel